CLINICAL TRIAL: NCT05675059
Title: Support Through Remote Observation and Nutrition Guidance (STRONG) Program for Pancreatic Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pancreatic Cancer Action Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-22082
Record Dates: First submitted 2022-12-09; First posted 2023-01-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Referral and Consultation; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: STRONG Intervention (Active Comparator): The STRONG program includes consultation with a Moffit dietician, logging intake of food daily into a food diary with a Fitbit smartphone app, and completing questionnaires.
  Interventions: Behavioral: Consultations with Moffitt Dietician; Behavioral: Daily Food Intake Diary with Fitbit Smartphone application; Behavioral: Questionnaires
- Group 2: Usual Care (Active Comparator): Participants will be referred to dieticians based on clinical discretion. Participants will also be asked to wear a Fitbit for 12 weeks to passively collect data on activity level.
  Interventions: Behavioral: Consultations with Moffitt Dietician; Behavioral: Daily Food Intake Diary with Fitbit Smartphone application; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Consultations with Moffitt Dietician — Participants will have an initial consultation and then biweekly follow-up visits (in-person or virtually) with a study dietician for 12 weeks.
Behavioral: Daily Food Intake Diary with Fitbit Smartphone application — Participants will keep a daily diary of food intake with a Fitbit smartphone app and wearing a Fitbit for 12 weeks.
Behavioral: Questionnaires — Participants will complete a questionnaire electronically at baseline and again at 4, 8, 12 and 16 weeks.

SUMMARY:
The purpose of the study is to assess the feasibility and participant satisfaction with the Support through Remote Observation and Nutrition Guidance (STRONG) program. The program provides enhanced dietician access and nutrition support for participants living with pancreatic cancer who are receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosed metastatic or newly recurrent pancreatic cancer or locally advanced pancreatic cancer
* Receiving chemotherapy under the guidance of Moffitt
* Able to speak and read English
* Able to provide informed consent

Exclusion Criteria:

* Documented or observable psychiatric or neurological disorder that would interfere with study participation (e.g., psychosis, active substance abuse).
* Undergoing concurrent treatment for a second primary GI cancer
* ECOG status of 2 or greater
* Use of parenteral or enteral nutrition
* Presence of malignant ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2025-11-22 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the STRONG Program | at 12 weeks
  Feasibility of the Support through Remote Observation and Nutrition Guidance (STRONG) program will be assessed using recruitment and retention rates, along with data completion rates.
Acceptability of the STRONG Program | at 16 weeks
  Acceptability of the STRONG Program measure uses 4 items to indicate participant satisfaction. The measure uses a scale of 0-5, 0 meaning the participant completely disagrees with the statements regarding intervention satisfaction and 5 indicating complete agreement with the statements regarding intervention satisfaction. The measure score ranges from 0-20 with 20 indicating the highest degree of satisfaction.
Participant adherence to the STRONG Program | Up to 90 days
  will be defined as ≥ 60% of patients will meet with a dietician for 4/6 dietician visits and ≥ 60% of patients will track daily food intake via a Fitbit.
Malnutrition: Significant Weight Loss | at 16 weeks
  Significant weight loss will be defined as a loss of >5% and >10% of body weight over the 16 week assessment period. Weight will be measured in kg.
Malnutrition: Low BMI | at 16 weeks
  Low BMI will be calculated by combining weight (kg) and height measurements (m²) and defined as <20kg/m² for adults < 70 years old and <22kg/m² for adults ≥ 70 years old over the 16 week assessment period.
Malnutrition: Low Skeletal Muscle Mass | at 16 weeks
  Low skeletal muscle mass will be calculated by estimating skeletal muscle index (SMI) by dividing the cross-sectional area of muscle in a single 'slice' from an abdominal CT scan (cm2) by stature (square of height in m²). Low SMI will be defined as ≤38.9 cm2/m2 for females and ≤55.4 for males over the 16 week assessment period.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Alishahi Tabriz, MD, PhD, MPH, Principal Investigator — Moffitt Cancer Center; Pamela Hodul, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Turner K, Kim DW, Gonzalez BD, Gore LR, Gurd E, Milano J, Riccardi D, Byrne M, Al-Jumayli M, de Castria TB, Laber DA, Hoffe S, Costello J, Robinson E, Chadha JS, Rajasekhara S, Hume E, Hagen R, Nguyen OT, Nardella N, Parker N, Carson TL, Tabriz AA, Hodul P. Support Through Remote Observation and Nutrition Guidance (STRONG), a digital health intervention to reduce malnutrition among pancreatic cancer patients: A study protocol for a pilot randomized controlled trial. Contemp Clin Trials Commun. 2024 Feb 23;38:101271. doi: 10.1016/j.conctc.2024.101271. eCollection 2024 Apr. PMID 38440777